CLINICAL TRIAL: NCT07058467
Title: Anterior Cruciate Ligaments: Studying Updates in neuroCognition After Knee Manipulation
Acronym: ACLs SUCK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-0824
Record Dates: First submitted 2025-06-18; First posted 2025-07-10 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-06

CONDITIONS: Anterior Cruciate Ligament (ACL) Tear; Anterior Cruciate Ligament Reconstruction Rehabilitation
Keywords: ACL; Anterior Cruciate Ligament; ACLR; Neurocognition
MeSH Terms: conditions — Lacerations

STUDY DESIGN:
Intervention Model Description: Single arm, pre-post cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Knee manipulation post ACLR (Experimental): This group, which comprises the entire cohort, will receive knee joint manipulations coinciding with grade III+ measures.
  Interventions: Other: Joint Manipulation

INTERVENTIONS:
Other: Joint Manipulation — A joint manipulation is defined as a manual treatment by a clinician that uses controlled force to improve joint function. For the purpose of this study, the terms manipulation and mobilization may be used interchangeably. The knee joint is specifically defined as the tibiofemoral articulation for the purpose of this study.
  All knee joint manipulation in this study will coincide with grade III or IV manipulations. This category coincides with evidence that mobilizations at or above grade III has the greatest impact on somatosensation and are most likely to produce a positive effect on neurocognitive function. Joint manipulation(s) will be delivered with a vector corresponding to the functional deficits found with manual joint palpation and will only occur with the involved ACLR knee. If both knees have experienced an ACL injury, the most recently injured knee will be manipulated.

SUMMARY:
This study will investigate whether knee joint manipulation can improve neurocognitive and neuromuscular performance in individuals with a history of anterior cruciate ligament reconstruction (ACLR). Recruitment will consist of 30 participants aged 18-35 who are 4 months to 5 years post-ACLR and demonstrate measurable reaction time delays. Using a within-subject pre-post design, participants will complete a battery of neurocognitive and neuromuscular assessments, including visuomotor reaction time and dual-task hop testing, before and after knee joint manipulation(s).

The main questions the investigators aim to address are:

Aim 1: Evaluate the feasibility, acceptability, and applicability of integrating knee joint manipulation into post-ACLR rehabilitation using the Implementation and Outcomes Framework.

Aim 2: Determine preliminary efficacy of knee joint manipulation on neurocognitive performance in individuals with ACLR.

ELIGIBILITY:
Inclusion Criteria:

* Provided informed consent prior to any study procedures that are performed.
* Are between the ages of 18 and 35.
* Have undergone ACLR surgery. All autograft and allograft types are accepted.
* Are 4-months to 10-years post-ACLR.
* Injured knee playing or training for sports (recreational or organized) or during physical activity.
* Have been cleared by a physician to return to activities and/or participate in this study.
* Are at least the minimally clinical important difference (MCID) above the normative reaction time average for our methods as established by previous literature in at least 1 reaction time task.

Exclusion Criteria:

* History of concussion in the past 3 months.
* The participant is pregnant.
* Have a neurological disorder, including epilepsy.
* Currently injured or have injured their lower extremity in the past 3 months.
* Had surgery on multiple ligaments when their ACL was injured.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Simple Reaction Time | Baseline and up to 90 minutes after completion of joint manipulation (intervention)
  Simple reaction time is the amount of time it takes for a person to respond to a single, known stimulus with a predefined response (ms). It is a basic measure of neuromuscular and cognitive processing speed. This is collected with the Senaptec Sensory Station.
Change in Lower Extremity Visuomotor Reaction Time | Baseline and up to 90 minutes after completion of joint manipulation (intervention)
  Visuomotor reaction time refers to the time it takes for an individual to see a visual stimulus and then generate a coordinated motor response to it (ms). It combines two processes: visual perception and motor execution. This is collected with the Fitlight system.
Mean Feasibility of Joint Manipulation Score | Baseline and up to 90 minutes after completion of joint manipulation (intervention)
  Collected with the Feasibility of Intervention Measure (FIM). Feasibility refers to how practical and achievable a study or project is in terms of its design, implementation, and resources. The FIM consists of four questions on a 5-point Likert scale ranging from 1 (completely disagree) to 5 (completely agree). The total score the four questions (4-20) will be averaged across all participants. Higher scores indicate greater feasibility. In this study, only patient perception is evaluated.
Mean Acceptability of Joint Manipulation Score | Baseline and up to 90 minutes after completion of joint manipulation (intervention)
  Collected with the Acceptability of Intervention Measure (AIM). Acceptability refers to how well a study's intervention, procedures, or overall design are perceived and tolerated by participants, clinicians, or other stakeholders. The AIM consists of four questions on a 5-point Likert scale ranging from 1 (completely disagree) to 5 (completely agree). The total score the four questions (4-20) will be averaged across all participants. Higher scores indicate greater acceptability. In this study, only patient perception is evaluated.
Mean Appropriateness of Joint Manipulation Score | Baseline and up to 90 minutes after completion of joint manipulation (intervention)
  Collected with the Intervention Appropriateness Measure (IAM). Appropriateness refers to the extent to which an intervention, method, or study design is suitable for the specific context, population, or problem being addressed. The IAM consists of four questions on a 5-point Likert scale ranging from 1 (completely disagree) to 5 (completely agree). The total score the four questions (4-20) will be averaged across all participants. Higher scores indicate greater appropriateness. This will only take into account the patient's response.

SECONDARY OUTCOMES:
Change in Mean Single Leg Hop Distance For Level 1 Neurocognitive Hop Test | Baseline and up to 90 minutes after completion of joint manipulation (intervention)
  Single leg hop distance (m) will be collected and averaged during three trials on both legs. The level 1 neurocognitive hop test consists of a Fitlight placed 3 meters directly in front of the participant to indicate when to jump and another light at the participant's feet. The Fitlight at the feet is used to measure the reaction time needed to jump once the "go" light activates. The target light will change colors in the order of red, yellow, then green and then the target "go" color. Once the participant lands, the distance hopped will be recorded.
Change in Mean Reaction Time For Level 1 Neurocognitive Hop Test | Baseline and up to 90 minutes after completion of joint manipulation (intervention)
  Single leg hop distance (m) will be collected and averaged during three trials on both legs. The level 1 neurocognitive hop test consists of a Fitlight placed 3 meters directly in front of the participant to indicate when to jump and another light at the participant's feet. The Fitlight at the feet is used to measure the reaction time needed to jump once the "go" light activates. The target light will change colors in the order of red, yellow, then green and then the target "go" color. Once the participant lands, the distance hopped will be recorded.
Change in Mean Single Leg Hop Distance For Level 2 Neurocognitive Hop Test | Baseline and up to 90 minutes after completion of joint manipulation (intervention)
  Single leg hop distance (m) will be collected and averaged during three trials on both legs. The level 2 neurocognitive hop test consists of Fitlights placed 3m directly in front and 45 degrees off center of the participant as the target lights. A Fitlight will also be placed at the participant's feet to measure reaction time off the start position. The left, center, or right light will be selected first via a counterbalancing method as the targeted light. The participant is not told which light will be the target light. The left Fitlight will change colors in the order of red, yellow, then green and then the target "go" color. Once the participant lands, the distance hopped will be recorded. All three directions (left, center, and right) are tested for each leg.
Change in Mean Reaction Time For Level 2 Neurocognitive Hop Test | Baseline and up to 90 minutes after completion of joint manipulation (intervention)
  Single leg hop distance (m) will be collected and averaged during three trials on both legs. The level 2 neurocognitive hop test consists of Fitlights placed 3m directly in front and 45 degrees off center of the participant as the target lights. A Fitlight will also be placed at the participant's feet to measure reaction time off the start position. The left, center, or right light will be selected first via a counterbalancing method as the targeted light. The participant is not told which light will be the target light. The left Fitlight will change colors in the order of red, yellow, then green and then the target "go" color. Once the participant lands, the distance hopped will be recorded. All three directions (left, center, and right) are tested for each leg.
Change in Mean Single Leg Hop Distance For Level 3 Neurocognitive Hop Test | Baseline and up to 90 minutes after completion of joint manipulation (intervention)
  Single leg hop distance (m) will be collected and averaged during three trials on both legs. The level 3 neurocognitive hop test consists of Fitlights placed 3m directly in front and 45 degrees off center of the participant as the target lights. For the level 3 test, a built in wait time with "no-go" colors flashing each second will be used. The wait time will be either 3, 4, or 5 seconds and is selected via counterbalancing without notifying the participant. The left Fitlight will change colors in the order of red, yellow, then green. Once the trial has started, the lights will flash different "no-go" colors once per second until the determined wait time has elapsed. One randomly selected light will change to the "go" color while the other lights will be a highly contrasted "no-go" color. Once the participant lands, the distance hopped will be recorded. All three added wait times are tested for each leg.
Change in Mean Reaction Time For Level 3 Neurocognitive Hop Test | Baseline and up to 90 minutes after completion of joint manipulation (intervention)
  Single leg hop distance (m) will be collected and averaged during three trials on both legs. The level 3 neurocognitive hop test consists of Fitlights placed 3m directly in front and 45 degrees off center of the participant as the target lights. A Fitlight will also be placed at the participant's feet to measure reaction time off the start position. For the level 3 test, a built in wait time with "no-go" colors flashing each second will be used. The wait time will be either 3, 4, or 5 seconds and is selected via counterbalancing without notifying the participant. The left Fitlight will change colors in the order of red, yellow, then green. Once the trial has started, the lights will flash different "no-go" colors once per second until the determined wait time has elapsed. One randomly selected light will change to the "go" color while the other lights will be a highly contrasted "no-go" color. All three added wait times are tested for each leg.

CONTACTS AND LOCATIONS:
Overall Officials: Shelby Baez, PhD, ATC, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 and continuing for 36 months following publication.
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.